CLINICAL TRIAL: NCT02919761
Title: A Multicenter, 2 Part Study to Assess the Efficacy and Safety of Acthar Gel in Subjects With Rheumatoid Arthritis With Persistently Active Disease Despite Dual-DMARD Treatment
Brief Title: Safety and Effectiveness of Acthar Gel in Participants With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MNK14294063
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Arthritis, Rheumatoid
Keywords: Persistent disease activity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Intervention Model Description: Part 1: Single Group; Part 2: Parallel
Who Masked: Participant, Investigator
Masking Description: Part 1: Open Label ; Part 2: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: All Enrolled Participants (Experimental): All participants receive Acthar Gel 1 mL twice weekly for 12 weeks
  Interventions: Drug: Acthar Gel
- Part 2: Acthar Gel (Experimental): Participants receive Acthar Gel 1 mL twice weekly for an additional 12 weeks
  Interventions: Drug: Acthar Gel
- Part 2: Placebo (Placebo Comparator): Participants receive Placebo 1 mL twice weekly for an additional 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acthar Gel — 80 Units Acthar Gel per 1 mL for subcutaneous injection
  Other Names: Acthar; H.P. Acthar Gel
  Arms: Part 1: All Enrolled Participants; Part 2: Acthar Gel
Drug: Placebo — Matching placebo 1 mL for subcutaneous injection
  Other Names: Matching Placebo
  Arms: Part 2: Placebo

SUMMARY:
This is a 2-part study to examine the effect of Acthar Gel in adult participants with rheumatoid arthritis (RA) with persistently active disease even after receiving two other treatments intended to modify the disease.

Part 1 is an Open Label Period in which all eligible participants receive Acthar Gel for 12 weeks. After these 12 weeks of treatment with Acthar Gel, participants will be evaluated for treatment response using the DAS28-ESR.

Participants who have achieved low disease activity (LDA) will enter a double-blind randomized maintenance period (Part 2) and be randomized in a 1:1 ratio to receive either Acthar Gel or matching placebo for an additional 12 weeks.

A single participant might be involved in the trial for as many as 32 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or nonpregnant, nonlactating female subjects
* Meets criteria for definite rheumatoid arthritis as defined by 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification at screening
* Has active disease defined as a score of >3.2 on DAS28-ESR prior to study drug administration despite dual-DMARD treatment
* Is on a stable dose of ≤ 20 mg per week of methotrexate for at least 8 weeks AND a stable dose of an allowed DMARD for at least 24 weeks prior to the screening visit
* May also be on a stable dose of 10 mg or less of prednisone or other the dose equivalent of another corticosteroid for 4 weeks prior to study drug administration

Exclusion Criteria:

* Has current rheumatoid disease or inflammatory joint disease other than RA
* Has any history of use of adrenocorticotropic hormone (ACTH) for the treatment of RA
* Has taken B-cell mediated therapies in the 6 months prior to screening
* Has hepatitis B, hepatitis C, history of tuberculosis (TB) or other contraindication as per the United States (US) Prescribing Information for Acthar
* Has history of Type 1 or Type 2 diabetes
* Has any clinically significant infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2016-11-07 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2019-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team Leader, Study Director — Mallinckrodt Pharmaceutical
Locations (59):
- United States (30):
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Orthopedic Research Institute, Boynton Beach, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - Southeastern Integrated Medical, PL, d/b/a Florida Medical Research, Gainesville, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Homestead Associates in Research, Homestead, Florida
  - Pharmax Research Clinic, Miami, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Omega Research Consultants-DeBary, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Arthritis & Rheumatology of Georgia, PC, Atlanta, Georgia
  - Arthritis Research and Treatment Center, Stockbridge, Georgia
  - Arthritis and Diabetes Clinic, Inc., Monroe, Louisiana
  - June DO, PC, Lansing, Michigan
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - DJL Clinical Research, Charlotte, North Carolina
  - Columbia Arthritis Center, Columbia, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Ramesh C. Gupta, MD, Memphis, Tennessee
  - Northwest Med Care, Cypress, Texas
  - Rheumatic Disease Clinical Research Center, Houston, Texas
  - Accurate Clinical Research, Houston, Texas
  - Laila Hassan, MD, PA, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Southwest Rheumatology Research, Mesquite, Texas
  - Sun Research Institute, San Antonio, Texas
- Argentina (4):
  - Aprillus Asistencia e Investigación, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - DIM Clínica Privada, Ramos Mejía, Buenos Aires
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Centro Polivalente de Asistencia e Investigación Clínica CER San Juan, San Juan
- Mexico (18):
  - Centro de Investigacion del Noroeste, S.C., Tijuana, Estado de Baja California
  - Antiguo Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad, Guadalajara, Jalisco
  - Investigacion Biomedica para el Desarrollo de Farmacos S.A. de C.V., Zapopan, Jalisco
  - Hospital De Jesus, Mexico City, Mexico City
  - Consultorio de Reumatología, Mexico City, Mexico City
  - Consultorio Privado del Dr. Miguel Cortes Hernandez, Cuernavaca, Morelos
  - Hospital Universitario Dr. José Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro de Estudios Clínicos y Especialidades Médicas, Monterrey, Nuevo León
  - Centro de Alta Especialidad en Reumatologia e Investigación del Potosí, San Luis Potosí City, San Luís Potosí
  - Centro Especializado en Investigación Clínica, Boca del Río, Veracruz
  - Centro Peninsular de Investigacion Clinica S.C.P., Mérida, Yucatán
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Phylasis Clinicas Research S de RL de CV, Estado de México
  - SMIQ, Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí, S.C., San Luis Potosí City
  - INBIOMEDYC Toluca, Toluca
  - Unidad de Enfermedades Reumaticas y Cronico Degenerativas, Torreón
- Peru (6):
  - Clinica Santa Monica, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - ABK Reuma S.R.L. - Medicentro Biociencias, Pueblo Libre
  - Clinica Vesalio, San Borja
  - Hospital de Apoyo Maria Auxiliadora, San Juán de Miraflores
  - Clínica Médica Cayetano Heredia, San Martín de Porres
- Mindful Medical Research, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fleischmann R, Furst DE. Safety of repository corticotropin injection as an adjunctive therapy for the treatment of rheumatoid arthritis. Expert Opin Drug Saf. 2020 Aug;19(8):935-944. doi: 10.1080/14740338.2020.1779219. Epub 2020 Jun 16. PMID 32497440
- [Derived] Fleischmann R, Furst DE, Connolly-Strong E, Liu J, Zhu J, Brasington R. Repository Corticotropin Injection for Active Rheumatoid Arthritis Despite Aggressive Treatment: A Randomized Controlled Withdrawal Trial. Rheumatol Ther. 2020 Jun;7(2):327-344. doi: 10.1007/s40744-020-00199-3. Epub 2020 Mar 17. PMID 32185745

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 259 patients were recruited at 80 study centers globally for Part 1. Of those participants, 77 were randomized to receive Acthar and 77 were randomized to receive Placebo for an additional 12 weeks, which was Part 2.
Pre-assignment Details: All participants enrolled in Part 1
Groups:
- All Enrolled Participants: All participants who enrolled in the trial
- Part 2: Acthar Gel: Participants receive 1 mL Acthar Gel twice weekly during Part 2, from Week 12 through Week 24
- Part 2: Placebo: Participants receive 1 mL placebo twice weekly during Part 2, from Week 12 through Week 24
Period: Part 1: Open Label
Arm/Group | All Enrolled Participants | Part 2: Acthar Gel | Part 2: Placebo
Started | 259 | 0 (Part 2 Blinded groups were not evaluated as such during Part 1) | 0
mITT Population (All participants who received study drug and contributed efficacy data.) | 259 | 0 | 0
Safety Population (All participants who received study drug.) | 259 | 0 | 0
Per Protocol Population (All participants who completed the Part 1 of the study without major protocol deviation.) | 236 | 0 | 0
Completed | 235 | 0 | 0
Not Completed | 24 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Met withdrawal criteria | 5 | 0 | 0
Not completed — Did Not Achieve Lda At Week 12 | 2 | 0 | 0
Not completed — Dose Greater Than 20mg/Week | 1 | 0 | 0
Not completed — did not meet inclusion criteria 8 | 1 | 0 | 0
Not completed — Termination by Sponsor | 1 | 0 | 0
Period: Part 2: Double-blind
Arm/Group | All Enrolled Participants | Part 2: Acthar Gel | Part 2: Placebo
Started | 0 (154 of the original Part 1 participants continued to Part 2, randomized to Acthar or placebo) | 77 (77 participants who completed Part 1 were to receive Acthar for an additional 12 weeks in Part 2) | 77 (77 participants who completed Part 1 were to receive placebo for an additional 12 weeks in Part 2)
Safety Population | 0 | 77 | 77
mITT Population | 0 | 77 | 76
Per Protocol Population | 0 | 76 | 73
Completed | 0 | 71 | 56
Not Completed | 0 | 6 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Met withdrawal criteria | 0 | 1 | 2
Not completed — Worsening of disease activity | 0 | 4 | 10
Not completed — Did not meet LDA at Week 16 | 0 | 0 | 1
Not completed — Did not meet LDA at Week 20 | 0 | 0 | 1
Not completed — Discontinued exclusion 16 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part 1: All Participants Enrolled: All participants who enrolled in the trial
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
Age, Continuous [Median (Full Range); unit: years] | 50 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 231
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 213
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 40
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 170
  More than one race | 0
  Unknown or Not Reported | 31

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Low Disease Activity (LDA) by Visit
Description: LDA is defined as DAS28 <3.2.
Time Frame: Baseline to Week 12
Population: modified Intent to Treat (mITT) Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
Participants
  at Baseline | 0
  at Week 4 | 17
  at Week 8 | 37
  at Week 12 | 163
Statistical Analysis 1: Comparison: Part 1: All Participants Enrolled; Test type: Other; p = 0.242, One-sample binomial test — At Week 4
Statistical Analysis 2: Comparison: Part 1: All Participants Enrolled; Test type: Other; p < 0.0001, One-sample binomial test — At Week 8
Statistical Analysis 3: Comparison: Part 1: All Participants Enrolled; Test type: Other; p < 0.0001, One-sample binomial test

2. Primary Outcome: Part 2: Number of Participants Who Maintained Low Disease Activity by Visit
Description: Low disease activity is defined as DAS28 <3.2.
Time Frame: Week 12 to Week 24
Population: mITT Population
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: Placebo: Participants receive Placebo 1 mL twice weekly during Part 2, from Week 12 through week 24
- Part 2: Acthar Gel: Participants receive Acthar Gel 1 mL twice weekly during Part 2, from Week 12 through Week 24
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 77 | 76
Participants
  at Week 12 | 77 | 75
  at Week 16 | 58 | 53
  at Week 20 | 61 | 48
  at Week 24 | 47 | 32
Statistical Analysis 1: Comparison: Part 2: Placebo vs Part 2: Acthar Gel; Test type: Other; p = 0.313, Pearson's Chi-square test — Comparison at Week 12
Statistical Analysis 2: Comparison: Part 2: Placebo vs Part 2: Acthar Gel; Test type: Other; p = 0.439, Pearson's Chi-square test — Comparison at Week 16
Statistical Analysis 3: Comparison: Part 2: Placebo vs Part 2: Acthar Gel; Test type: Other; p = 0.028, Pearson's Chi-square test — Comparison at Week 20
Statistical Analysis 4: Comparison: Part 2: Placebo vs Part 2: Acthar Gel; Test type: Other; p = 0.019, Pearson's Chi-square test — Comparison at Week 24

3. Secondary Outcome: Part 1: Swollen Joint Count by Visit
Description: The investigator counts the number of swollen joints used to calculate the Disease Activity Score (DAS28-ESR, DAS28)
  The DAS28 is a composite score derived from the following assessments:
  * Swollen Joint Count
  * Tender Joint Count
  * Patient's Global Health
  * Erythrocyte Sedimentation Rate
Time Frame: Baseline to Week 12
Population: mITT
Measure: Mean (Standard Deviation); unit: Count of swollen joints
Units Other Than Participants: Joints
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
Number analyzed (Joints) | 28
Count of swollen joints
  at Baseline | 10.9 (5.37)
  at Week 4 | 5.6 (4.88)
  at Week 8 | 4.0 (4.36)
  at Week 12: number analyzed (Participants) | 258
  at Week 12 | 2.8 (4.26)

4. Secondary Outcome: Part 2: Swollen Joint Count by Visit During Part 2
Description: The investigator counts the number of swollen joints used to calculate the Disease Activity Score (DAS28-ESR/DAS28)
  The DAS28 is a composite score derived from the following assessments:
  * Swollen Joint Count
  * Tender Joint Count
  * Patient's Global Health
  * Erythrocyte Sedimentation Rate
Time Frame: Baseline, Week 12 to Week 24
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Count of swollen joints
Units Other Than Participants: Joints
Groups:
- Part 2: Placebo: Participants receive Placebo during Part 2
- Part 2: Acthar Gel: Participants who receive Acthar Gel during Part 2
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 76 | 77
Number analyzed (Joints) | 28 | 28
Count of swollen joints
  at Baseline | 10.1 (4.87) | 9.7 (4.32)
  at Week 12 | 0.9 (1.09) | 0.9 (1.03)
  at Week 16 | 1.7 (3.08) | 1.1 (1.31)
  at Week 20 | 1.9 (3.62) | 0.9 (1.19)
  at Week 24 | 2.3 (3.71) | 1.5 (2.29)

5. Secondary Outcome: Part 1: Tender Joint Count by Visit
Description: The investigator counts the number of tender joints used to calculate the Disease Activity Score (DAS28-ESR, DAS28)
  The DAS28 is a composite score derived from the following assessments:
  * Swollen Joint Count
  * Tender Joint Count
  * Patient's Global Health
  * Erythrocyte Sedimentation Rate
Time Frame: Baseline to Week 12
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Count of Tender Joints
Units Other Than Participants: Joints
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
Number analyzed (Joints) | 28
Count of Tender Joints
  at Baseline | 14.7 (7.08)
  at Week 4 | 7.7 (6.39)
  at Week 8 | 5.7 (5.93)
  at Week 12: number analyzed (Participants) | 258
  at Week 12 | 3.9 (5.69)

6. Secondary Outcome: Part 2: Tender Joint Count by Visit
Description: as for outcome 5
Time Frame: Baseline, Week 12 to Week 24
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Count of Tender Joints
Units Other Than Participants: Joints
Groups:
- Part 2: Placebo: Participants who receive Placebo during Part 2
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 76 | 77
Number analyzed (Joints) | 28 | 28
Count of Tender Joints
  at Baseline | 13.5 (7.24) | 13.5 (6.41)
  at Week 12 | 1.5 (1.33) | 1.4 (1.24)
  at Week 16 | 2.6 (3.96) | 1.6 (1.47)
  at Week 20 | 2.7 (4.36) | 1.5 (1.67)
  at Week 24 | 3.1 (4.46) | 2.4 (4.29)

7. Secondary Outcome: Part 1: Patient-Reported General Health by Visit
Description: Participants rate their general health on a 100 mm visual analogue scale (VAS), where 0=best general health and 100=worst general health.
  A lower score indicates better general health.
Time Frame: Baseline to Week 12
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
mm
  at Baseline | 59.8 (20.02)
  at Week 4 | 45.1 (23.15)
  at Week 8 | 37.8 (22.95)
  at Week 12 | 27.0 (22.18)

8. Secondary Outcome: Part 2: Patient-Reported General Health by Visit
Description: as for outcome 7
Time Frame: Baseline, Week 12 to Week 24
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 76 | 77
mm
  at Baseline | 13.5 (7.24) | 13.5 (6.41)
  at Week 12 | 15.4 (14.47) | 18.8 (14.34)
  at Week 16 | 17.2 (18.16) | 19.6 (17.98)
  at Week 20 | 18.5 (20.14) | 17.9 (16.04)
  at Week 24 | 21.4 (22.56) | 21.3 (21.28)

9. Secondary Outcome: Part 1: Erythrocyte Sedimentation Rate (ESR) by Visit
Description: The ESR is the rate at which red blood cells (in whole blood that has not clotted) fall to the bottom of the tube over a period of one hour.
  The clear liquid above the red blood cells is measured in millimeters after one hour (mm/hr).
  The normal range for ESR results is 1-13 mm/hr for males and 1/20 mm/hr for females.
  The ESR is a common test for inflammation and used to derive the DAS28.
  The DAS28 is a composite score derived from the following assessments:
  * Swollen Joint Count
  * Tender Joint Count
  * Patient's Global Health
  * Erythrocyte Sedimentation Rate
Time Frame: Baseline to Week 12
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
mm/hr
  at Baseline | 43.6 (24.77)
  at Week 4 | 35.4 (23.04)
  at Week 8 | 30.6 (21.24)
  at Week 12 | 24.0 (21.54)

10. Secondary Outcome: Part 2: Erythrocyte Sedimentation Rate (ESR) by Visit
Description: as for outcome 9
Time Frame: Baseline, Week 12 to Week 24
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 76 | 77
mm/hr
  at Baseline | 42.2 (23.05) | 40.3 (21.47)
  at Week 12 | 15.2 (12.669) | 15.8 (12.21)
  at Week 16 | 19.6 (14.62) | 17.7 (14.42)
  at Week 20 | 22.0 (17.75) | 17.5 (13.67)
  at Week 24 | 25.1 (18.81) | 23.1 (16.56)

11. Secondary Outcome: Part 1: Patient's Global Assessment of Pain by Visit
Description: Patients rate their pain on a 100 mm VAS, where 0=no pain and 100=pain as bad as it could be. Higher scores indicate more pain.
Time Frame: Baseline to Week 12
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
mm
  at Baseline | 64.9 (20.36)
  at Week 4 | 44.1 (23.78)
  at Week 8 | 37.3 (22.92)
  at Week 12 | 27.5 (23.02)

12. Secondary Outcome: Part 2: Patient's Global Assessment of Pain by Visit
Description: as for outcome 11
Time Frame: Baseline, Week 12 to Week 24
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 76 | 77
mm
  at Baseline | 62.8 (21.02) | 65.7 (18.65)
  at Week 12 | 17.0 (16.00) | 18.9 (16.64)
  at Week 16 | 21.6 (21.72) | 22.1 (20.77)
  at Week 20 | 20.0 (20.21) | 19.8 (16.23)
  at Week 24 | 22.1 (20.50) | 21.8 (19.70)

13. Secondary Outcome: Part 1: Physician's Global Assessment of Disease Activities by Visit
Description: The physician rates the participant's disease activity on a 100 mm visual analogue scale, where 0=very good and 100=very bad. Lower scores indicate improvement.
Time Frame: Baseline to Week 12
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 1: All Participants Enrolled
Number analyzed (Participants) | 259
mm
  at Baseline | 64.3 (14.93)
  at Week 4 | 36.1 (18.90)
  at Week 8 | 29.0 (18.92)
  at Week 12 | 21.0 (19.49)

14. Secondary Outcome: Part 2: Physician's Global Assessment of Disease Activities by Visit
Description: as for outcome 13
Time Frame: Week 12 to Week 24
Population: mITT Population
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part 2: Placebo | Part 2: Acthar Gel
Number analyzed (Participants) | 77 | 77
mm
  at Week 12 | 11.5 (8.91) | 12.9 (11.49)
  at Week 16 | 15.5 (15.57) | 13.3 (13.78)
  at Week 20 | 15.9 (16.25) | 12.4 (8.61)
  at Week 24 | 17.8 (18.12) | 15.2 (16.84)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected during an active treatment period of 24 weeks, and a follow-up visit of 28 (± 2) days after last dose of study drug
Groups:
- Part 1: All Participants Enrolled: All participants enrolled in the trial with AEs during Part 1
- Part 2: Placebo: Participants who received Placebo in Part 2 with AEs during Part 2
- Part 2: Acthar Gel: Participants who received Acthar Gel in Part 2 with AEs during Part 2
Arm/Group | Part 1: All Participants Enrolled | Part 2: Placebo | Part 2: Acthar Gel
All-Cause Mortality (participants affected / at risk) | 0/259 | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 3/259 | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 26/259 | 26/77 | 22/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: All Participants Enrolled (N=259) | Part 2: Placebo (N=77) | Part 2: Acthar Gel (N=77)
Chest pain (General disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: All Participants Enrolled (N=259) | Part 2: Placebo (N=77) | Part 2: Acthar Gel (N=77)
Urinary tract infection (Infections and infestations) | 10 | 3 | 2
Pharyngitis (Infections and infestations) | 7 | 0 | 0
Headache (Nervous system disorders) | 9 | 5 | 5
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 0
Rhinitis (Infections and infestations) | 0 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Glycosylated haemoglobin increased (Investigations) | 0 | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 2
Hypertension (Vascular disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT02919761/Prot_SAP_000.pdf